CLINICAL TRIAL: NCT04658329
Title: Cohorte ANRS CO5 "Cohorte Nationale VIH2"
Brief Title: Cohorte Nationale VIH-2
Acronym: ANRS CO VIH2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS CO5 VIH-2
Record Dates: First submitted 2020-08-05; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: HIV-2 Infection
Keywords: virus; HIV; cohort
MeSH Terms: conditions — Virus Diseases | interventions — Anti-Retroviral Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antiretroviral — Study the response to antiretroviral treatment (clinical, immuno-virological) and contribute to the identification of the antiretroviral strategies and combinations most suited to the particularities of the infection.

SUMMARY:
The HIV2 study is an open cohort of prospective, multicentric, national observation. The main objective is to study HIV-2 infection in adult patients followed in France.

DETAILED DESCRIPTION:
The secondary objectives are :

* Describe the epidemiological and clinical characteristics of participants infected with HIV-2, and the immuno-virological characteristics of the infection.
* To study the clinical and immunological progression of HIV-2 infection and the prognostic factors of this evolution.
* Study the response to antiretroviral treatment (clinical, immuno-virological) and contribute to the identification of the antiretroviral strategies and combinations most suited to the particularities of the infection.
* Allow an evaluation of the care practices of participants followed in French hospitals
* Provide a bank of clinical-biological data and samples allowing the performance of virological and / or immunological studies on HIV-2 infection.

The follow-up of the participants is different according to the therapeutic status of the participants, naive of antiretroviral treatment or already treated with antiretrovirals.

ELIGIBILITY:
Inclusion Criteria:

* HIV-2 infection only, diagnosed by ELISA, confirmed by Western-Blot test,
* Follow-up in consultation or hospitalization in one of the investigating centers,
* Age greater than or equal to 18 years,
* Prolonged follow-up possible, residence in France planned for at least one year,
* Consent to participate,
* Long-term medical care possible for the participant, or by medical aid (AME), or declaration of obtaining AME at the time of inclusion.

Exclusion Criteria:

* HIV-1 infection
* Double HIV-1 + HIV-2 seropositivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-2 infection only followed in consultation or hospitalization in one of the participating centers in France
Sampling Method: Non-Probability Sample
Enrollment: 1185 (Estimated)
Dates: Start 1994-01-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Study HIV-2 infection rate in adult patients followed in France | At the baseline

SECONDARY OUTCOMES:
The clinical progression of patients infected HIV-2 evaluate by samples: biological examinations | Up to 25 years
  Every 6 months
The epidemiological parameters and progression of patients infected with HIV-2 evaluate by a questionnaire | Up to 25 years
  Every 6 months
The rate of immuno-virological charge of the infection evaluate by serology samples | Up to 25 years
  Every 6 months
Pourcentage of patient with HIV-2 | Up to 25 years
  The prognostic factors of patient evolution are evaluate by biological samples
Pourcentage of response to antiretroviral treatment evaluate by serology samples | Up to 25 years
Pourcentage of good management practices of patients followed in French hospitals evaluate by results | Up to 25 years
  During the procedure

CONTACTS AND LOCATIONS:
Overall Officials: François Dabis, Pr, MD, Study Director — ANRS, Emerging Infectious Diseases
Locations (29):
- France (29):
  - Centre hospitalier Victor Dupouy, Argenteuil
  - Avicenne, Bobigny
  - Hôpital Saint André, Bordeaux
  - Service de Medecine Interne Hopital Antoine Beclere, Clamart
  - Hôpital Louis Mourier, Colombes
  - Hôpital Sud Francilien, Corbeil-Essonnes
  - Hôpital Henri Mondor, Créteil
  - Service de Médecine interne - Centre Hospitalier Intercommunal, Créteil
  - Hôpital Edouard Herriot, Lyon
  - Hôpital de La Croix Rousse, Lyon
  - Centre Hospitalier François Quesnay, Mantes-la-Jolie
  - Hôpital Gui de Chaudiac, Montpellier
  - Hôpital de l'Hotel Dieu, Nantes
  - Hôpital Saint Louis, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital la Pitié Salpétrière, Paris
  - Service de Medecine Interne Hopital Cochin, Paris
  - Hôpital Bichat - Claude Bernard, Paris
  - Hôpital Tenon, Paris
  - Hôpital Hôtel Dieu, Paris
  - Hôpital Lariboisière, Paris
  - Hopital du Kremlin Bicêtre Service de médecine interne, Paris
  - Centre Hospitalier René Dubos, Pontoise
  - Hôpital Pontchaillou, Rennes
  - Hôpital Delafontaine, Saint-Denis
  - CHI Poissy Saint Germain en Laye, Saint-Germain-en-Laye
  - Hôpital Bretonneau - Service des Maladies Infectieuses, Tours
  - Hôpital André Mignot, Versailles
  - CHI Villeneuve Saint Georges, Villeneuve-Saint-Georges